CLINICAL TRIAL: NCT05233774
Title: Lomecel-B Effects on Alzheimer's Disease: A Randomized, Double-Blinded, Placebo-Controlled Phase 2a Trial
Brief Title: Lomecel-B Effects on Alzheimer's Disease
Acronym: CLEARMIND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-007-01
Record Dates: First submitted 2021-12-16; First posted 2022-02-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mild Alzheimer's Disease

STUDY DESIGN:
Intervention Model Description: The study consists of 4 study arms of 12 patients each.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Group 1 will receive four infusions of Placebo on Day 0, Week 4, Week 8, and Week 12.
  Interventions: Other: Placebo
- Lomecel-B Dose 1 (Experimental): Group 2 will receive an infusion of Lomecel-B at a dose of 25 x 10^6 cells (25M) on Day 0, followed by Placebo infusions at Week 4, Week 8, and Week 12.
  Interventions: Drug: Allogeneic MSC
- Lomecel-B Dose 2 (Experimental): Group 3 will receive four infusions of 25M Lomecel-B on Day 0, Week 4, Week 8, and Week 12.
  Interventions: Drug: Allogeneic MSC
- Lomecel-B Dose 3 (Experimental): Group 4 will receive four infusions of Lomecel-B at a dose of 100 x 10^6 cells (100M) on Day 0, Week 4, Week 8, and Week 12.
  Interventions: Drug: Allogeneic MSC

INTERVENTIONS:
Drug: Allogeneic MSC — An allogeneic bone marrow-derived medicinal signaling cell (MSC) formulation
  Arms: Lomecel-B Dose 1; Lomecel-B Dose 2; Lomecel-B Dose 3
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Dementia resulting from AD is associated with vascular function decline and involves a pro-inflammatory state. In our Phase 1 trial, Lomecel-B treatment met the primary safety endpoint, with no safety concerns, and showed potential to improve clinical assessments. Mechanistically, Lomecel-B treated subjects had higher serum concentrations of pro-vascular and anti-inflammatory biomarkers relative to placebo. This trial builds upon those preliminary Phase 1 results, and is designed to evaluate the safety profile of multiple infusions of Lomecel-B, and to investigate provisional efficacy of single dosing versus multiple dosing of Lomecel-B on cognitive function and biomarkers in AD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Be 60 - 85 years of age at signing of the Informed Consent Form.
* Clinical diagnosis of mild Alzheimer's disease in accordance with the NIA-AA criteria at the time of enrollment.
* MMSE score of 19 - 23.
* Body weight of 40 - 150 kg.
* Has an adult caregiver who meets all of the following criteria.

  1. Provides written informed consent to participate on the trial (reporting on patient observations).
  2. Either lives with the patient, or sees the patient for at least 2 hours/day for at least 3 days/week.
  3. Is willing and able to participate in the study, and agrees to accompany the patient to each study visit.
  4. Is able to read, understand, and speak the designated language at the study site.
* Brain MRI consistent with AD.
* A PET scan using an FDA-approved tracer (e.g., AMYViD, Vizamyl, or Neuraceq) consistent with the diagnosis of AD. A prior positive PET scan will be allowed with Sponsor approval.
* Living in the community, includes assisted living facilities (but excluding long-term care nursing facilities).

Exclusion Criteria:

* Diagnosed with frontotemporal dementia (FTD), dementia due to Acquired Immunodeficiency Syndrome (AIDS), Creutzfeldt-Jakob disease (CJD), Lewy Bodies dementia (LBD), Progressive Supranuclear Palsy (PSP), multiple cerebral infarctions, or normal pressure hydrocephalus.
* Any other neurodegenerative disease.
* History of a seizure disorder.
* Evidence of: a prior macrohemorrhage; at least 4 cerebral microhemorrhages (regardless of anatomical location or diagnostic characterization as "possible" or "definite"); or at least 1 area of superficial siderosis.
* Unwillingness or inability to have MRIs scans (no contrasting agent will be used), or condition that contraindicates MRI, such as the presence metallic objects in the eyes, skin, or heart.
* Any conditions that contraindicates PET with a beta-amyloid tracer.
* Significant intestinal malabsorption surgery, e.g., gastric bypass.
* Serum B12 and/or folate levels below normal range.
* Clinically abnormal free T4 or thyroid-stimulating hormone (TSH).
* Resting blood oxygen saturation <93%.
* Resting systolic blood pressure >180 mm Hg, or diastolic blood pressure >110 mm Hg.
* Regularly (> 4 weeks) using high-doses of corticosteroids or other steroidal anti-inflammatory medication (e.g., Prednisone) on a regular basis, with the exception of steroidal nasal sprays, asthma inhalers, topical steroids, and hormonal-replacement therapy.
* Regularly (> 4 weeks) using anti-cytokine antibody or targeting therapy, e.g., anti-TNF-α.
* Be an organ transplant recipient, or have active or expected future listing for any organ/tissue transplant while scheduled to be on trial, except for corneal, bone, skin, ligament, or tendon.
* Diagnosed with malignancy within the past 2 years, with the exception of curatively treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ, or cervical carcinoma.
* Known hypersensitivity to dimethyl sulfoxide (DMSO).
* Test positive for hepatitis B virus surface antigen, viremic hepatitis C virus, HIV, or syphilis.
* Any condition that is projected to limited life expectancy to < 12 months.
* Be pregnant, nursing, or of childbearing potential while not practicing effective contraception.
* Be currently participating in any other investigational therapeutic or device trial, or have participated within one within the previous 30 days to screening, or in the opinion of the investigator, the patient should be excluded for such participation within the past 5 years.
* In the opinion of the investigator, the patient has any other illness or condition that: may compromise the participant's safety, compliance, or ability to successfully complete the study; may compromise the validity of the study; or otherwise should exclude the participant from enrollment.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint 1: Safety - SAEs and AEs | 41 weeks
  To demonstrate that Lomecel-B infusions do not trigger the pre-specified stopping rules.
  Additional safety will be acquired throughout the study as follows: Incidence of all AEs and SAEs over the course of the trial.
Primary Endpoint 2: Safety - Imaging | 41 weeks
  To demonstrate that Lomecel-B infusions do not trigger the pre-specified stopping rules.
  Additional safety will be acquired throughout the study as follows: Alzheimer's disease-related imaging abnormalities (ARIA) or clinically asymptomatic microhemorrhages as revealed by MRI.

SECONDARY OUTCOMES:
Secondary Endpoint 2: Efficacy- Change in the ADAS-cog-13 | 41 weeks
  Change from baseline in the ADAS-cog-13 in Lomecel-B-treated arms versus change in placebo.
Secondary Endpoint 3: Efficacy- Change in the MMSE | 41 weeks
  Change from baseline in the MMSE in Lomecel-B-treated arms versus change in placebo.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Visionary Investigators Network, Aventura, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Science Connections - Research Partner Group Multispecialty Group, Doral, Florida
  - Bruce W. Carter VA Medical Center, Miami, Florida
  - Miami Jewish Health, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Ivetmar Medical Group, Miami, Florida
  - Fusion Medical Research and Clinic, Miami, Florida
  - First Excellent Research Group, LLC, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Imic Inc., Palmetto Bay, Florida
  - Brain Matters Research, Stuart, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rash BG, Ramdas KN, Agafonova N, Naioti E, McClain-Moss L, Zainul Z, Varnado B, Peterson K, Brown M, Leal T, Kopcho S, Carballosa R, Patel P, Brody M, Herskowitz B, Fuquay A, Rodriguez S, Jacobson AF, Leon R, Pfeffer M, Schwartzbard JB, Botbyl J, Oliva AA Jr, Hare JM. Allogeneic mesenchymal stem cell therapy with laromestrocel in mild Alzheimer's disease: a randomized controlled phase 2a trial. Nat Med. 2025 Apr;31(4):1257-1266. doi: 10.1038/s41591-025-03559-0. Epub 2025 Mar 10. PMID 40065171